CLINICAL TRIAL: NCT05713474
Title: Micro-EMG: A Novel Multi-electrode System for Intramuscular Imaging of Human Motor Units
Brief Title: Micro-EMG: A Novel Multi-electrode System for Intramuscular Imaging
Status: Recruiting | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: uEMG; 280391 (Other: IRAS); 22-NS-0097 (Other: Ethics approval HRA)
Record Dates: First submitted 2023-01-12; First posted 2023-02-06 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Electromyography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy controls
  Interventions: Diagnostic Test: Diagnostic EMG exam with microEMG; Diagnostic Test: Conventional EMG
- Patients previously diagnosed with motor neurone disease
  Interventions: Diagnostic Test: Diagnostic EMG exam with microEMG; Diagnostic Test: Conventional EMG
- Patients previously diagnosed with sarcopenia
  Interventions: Diagnostic Test: Diagnostic EMG exam with microEMG; Diagnostic Test: Conventional EMG
- Patients previously diagnosed with post-polio syndrome
  Interventions: Diagnostic Test: Diagnostic EMG exam with microEMG; Diagnostic Test: Conventional EMG
- Patients previously diagnosed with myasthenia gravis
  Interventions: Diagnostic Test: Diagnostic EMG exam with microEMG; Diagnostic Test: Conventional EMG

INTERVENTIONS:
Diagnostic Test: Diagnostic EMG exam with microEMG — Diagnostic EMG exam with microEMG
Diagnostic Test: Conventional EMG — Diagnostic EMG exam with conventional EMG

SUMMARY:
The purpose of this small-scale exploratory study is to bridge the knowledge gap between the bench testing and the design of potential future confirmative studies. Identifying and evaluating MicroEMG measurement parameters in this exploratory manner is a necessary step to evaluate its usability and design, and determine whether the microEMG system may be suitable for in-house use after further confirmative testing.

DETAILED DESCRIPTION:
About this study We have developed a completely new multi-electrode electromyography system (MicroEMG) that we want to test in this study. It records muscle activity from multiple recording points in the muscle at once. We believe that this will increase the sensitivity of the technique in diagnosing muscle disease, reduce the time taken, and be more comfortable for patients. However, to prove whether this is the case we first need to understand the how the recorded signals of the new MicroEMG look like in different patient groups.

Background:

Why are we doing this study?

Electromyography (EMG) is an essential diagnostic test for nerve and muscle diseases. Cells in the muscle generate electric potentials when they are activated. This activity can be measured by the EMG. Based on those 'patterns', experts can detect medical abnormalities, such as muscle or nerve disorders. EMG involves inserting a thin metal needle electrode through the skin into a muscle. It records changes in the pattern of electrical signals produced by the muscle fibres. In conventional EMG only a single recording surface at the tip of the needle is used and therefore only small part of muscle can be examined.

We developed a new EMG device called MicroEMG. It uses a novel type of electrode that can examine the muscle in more detail. As it records activity from several different points at the muscle at once it can produce an electrical image (rather than an abstract signal). This way a large volume of muscle can be recorded simultaneously with less movement and discomfort for the patient.

What is the goal of this study?

Patients with a disease known to affect the nerves or the muscles typically would be tested with conventional EMG. Some diseases are linked to a specific 'diagnostic pattern' in the EMG that guides the specialist's diagnosis.

We do not know these pattern for MicroEMG yet. In this study we want to look at how measurements with the new MicroEMG look like in patients with neuromuscular disease. Each patient will undergo recordings from identical muscles using both conventional EMG and microEMG during a single visit. This will allow us to relate the electrical signal patterns in the muscle measured by MicroEMG to the known diagnostic pattern we typically see in conventional EMG. We will do this in both healthy and diseased muscles. Based on that we can determine which of these patterns may be suitable as potential diagnostic markers for the MicroEMG system.

We will also ask participants about their experience as a patient. It will give us a better understanding about how patients in our hospital may benefit from the new MicroEMG device in the future (after further confirmative research).

Who can participate?

In this study we want to look at how measurements with the new MicroEMG look like in patients with neuromuscular diseases - in particular, motor neurone disease, sarcopenia, post-polio syndrome, and myasthenia gravis. We also want to look at how those signals compare to signals measured in a healthy control group.

Participants will have a previously known diagnosis of any of the abovementioned diseases.

Not everyone is able to take part. Important reasons why one may not be able to take part include:

* Having a cardiac pacemaker or implanted defibrillator.
* Alternative neurological disorders.
* Lymphedema or dialysis fistula in the arms or legs.
* Taking clotting inhibitors or having a clotting disorder.

What does the study involve? What will I be asked to do?

Initial appointment

* We will ask participants to attend the Neurophysiology Department in Newcastle Hospitals NHS Trust.
* We will ask participants to fill out a data entry form (e.g. age, gender and contact details).
* We will ask participants basic questions about their health history to ensure they are able to take part.

Recording EMG

* We will perform 2 EMG exams, one with a conventional EMG needle that is normally used in our clinic. Another exam we will use the newly developed MicroEMG.
* We will ask participants to put their phone in flight mode (if possible) and lie on a couch.
* For each exam we will place a fine needle into in the muscles in the arms and shins (in total 5 different points). The insertion spots will be cleaned using alcohol beforehand.
* The EMG procedures are uncomfortable and can cause a similar amount of pain to having a vaccination. They may cause some temporary bruising to the skin but have no long-term effects.
* Each EMG exam will take approximately 30 minutes.
* At the end of each exam, we will ask participants to fill in a short questionnaire. This is to learn about their experience of the EMG exam, any discomfort, and any suggestions for improvement.
* We expect the entire procedure to not take longer than 2 hours.

What are the possible benefits of taking part?

* This study itself will not benefit participants. We expect the results of this study will help us decide us whether and how MicroEMG may be used as a diagnostic tool in our hospital in the future.
* We hope that this new system will help with the future diagnosis of diseases which damage the nerves and muscles. However, to prove this systematically we need to do more research.

What are the possible risks of taking part?

* The needle test (electromyography) is uncomfortable but has no long-term effects.
* In people with blood clotting abnormalities there is a small risk of bleeding inside the muscles. To avoid this, anyone with blood clotting problems will be excluded from the study as a precaution.
* To control risk of infection we clean the skin with alcohol before inserting the sterile needle. After use, the needle is safely disposed.
* In addition, our department has put in place extensive measures to ensure patient safety during the Covid-19 pandemic. These have been reviewed and approved by the hospital Infection Control Team.

Who monitors this study?

• The study is overseen by Newcastle Upon Tyne Hospitals NHS Foundation Trust (NuTH). It is a requirement that participant records in this research, together with any relevant medical records, be made available for scrutiny by monitors from NuTH. Their role is to check that research is properly conducted and the interests of those taking part are adequately protected. NIHR-BRC has provided funding for this study.

Who can I contact for further information? If you would like further information please contact Dr Roger Whittaker (0191 28 24578 or 0191 2083543) or Katrin Bangel (Katrin.Bangel[at]nhs.net)

ELIGIBILITY:
Inclusion Criteria:

* For each of the five groups, six participants will be recruited, adding up to a total of 30 participants.

Exclusion Criteria:

* cardiac pacemakers or defibrillator implants.
* alternative neurological disorders likely to affect the results of an EMG examination.
* lymphedema or dialysis fistula in the body region to be studied with EMG.
* patients taking clotting inhibitor (such as warfarin or direct oral anticoagulants).
* clotting disorder (such as haemophilia or low platelets).
* participants unable to consent in English where a translator is not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with neuromuscular diseases - in particular, motor neurone disease, sarcopenia, post-polio syndrome, and myasthenia gravis - as well as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
List of potential EMG parameters to inform future diagnostic marker evaluation studies. | 1 study day
  extracted from EEG recordings
Report of tested and potential vs. disregarded diagnostic markers for MicroEMG. | 1 study day
  extracted from EEG recordings

SECONDARY OUTCOMES:
Summary of health care and patient experience with MicroEMG system. | 1 study day
  questionnaire
Potential changes to the system or the examination procedure. | 1 study day
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Roger Whittaker, Principal Investigator — Newcastle University
Locations (1):
- RVI - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No